CLINICAL TRIAL: NCT04699916
Title: EEG-based Protocol to Guide Deep Sedation Decreases the Days of Mechanical Ventilation in Patients With SARS-CoV-2 Pneumonia: Randomized Clinical Trial
Brief Title: EEG-based Sedation Protocol for Patients on Mechanical Ventilation Due to SARS-CoV-2 Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Rodrigo Gutiérrez, Assistant Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 80320
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Sedation Complication; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Deep Sedation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Usual care) (No Intervention): Sedation will be guided with a standard protocol based on Sedation Agitation Scale already implemented in the Intensive Care Unit
- EEG-based sedation protocol (Experimental): Sedation will be guided using a protocol based on 2 parameters from the EEG: Suppression Rate and Spectral Edge Frequency
  Interventions: Other: EEG based protocol for deep sedation

INTERVENTIONS:
Other: EEG based protocol for deep sedation — Protocol established to guide sedation drug dosification to maintain the patient with a Suppression Rate (SR) less than 1% and a Spectral Edge Frequency 95 over 10 Hz
  Arms: EEG-based sedation protocol

SUMMARY:
Deep sedation in patients with COVID-19 may be challenging in many aspects. The use of an EEG-based protocol to guide deep sedation may be useful in this particular population, considering their unusually high sedation requirements.

In the present trial, we aim to evaluate an EEG-based protocol to guide deep sedation in patients with COVID19, using to EEG derived parameters that are displayed in the BIS monitor: Suppression Rate and Spectral Edge Frequency.

The protocol is designed to both minimize the suppression rate along with maintaining a spectral edge frequency over 10 Hz. The use of this protocol may reduce the amount of sedatives administered and, therefore, diminish the time needed for the weaning process.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* COVID-19 patient requiring mechanical ventilation

Exclusion Criteria:

* Contraindication to receive propofol or fentanyl
* Chronic Liver Disease Child C
* End-Stage Kidney Chronic Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-05-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Ventilator Free Days | Day 30
  Number of days in which the patient is both alive and out of the invasive mechanical ventilator

SECONDARY OUTCOMES:
Plasma propofol concentration | Day 5
  Plasma propofol concentration measure with HPLC
Total administered dose of propofol | Day 5
  Accumulated Dose of propofol administered in mg/kg
Total administered dose of Fentanyl | Day 5
  Accumulated Dose of fentanyl administered in mcg/kg
Total administered dose of Norepinephrine | Day 5
  Accumulated Dose of norepinephrine administered in mcg/kg
Propofol-Related Infusion Syndrome (PRIS) Incidence | Day 30
  Diagnosis of PRIS
Accidental extubation | Day 30
  Occurrence of a non-planned extubation
Delirium Incidence | Day 30
  Diagnosis of delirium with CAM-ICU
ICU length of stay | Day 30
  Nights spent in the ICU
Hospital length of stay | Day 90
  Nights spent in the ICU
Mortality | Day 30
  Mortality
Success of the first weaning trial | Day 30
  Patients who succeed the first weaning trial and are extubated without difficulty, according to the WIND trial definition

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico de la Universidad de Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID 32227758
- [Background] Kollef MH, Levy NT, Ahrens TS, Schaiff R, Prentice D, Sherman G. The use of continuous i.v. sedation is associated with prolongation of mechanical ventilation. Chest. 1998 Aug;114(2):541-8. doi: 10.1378/chest.114.2.541. PMID 9726743
- [Background] Hanidziar D, Bittner EA. Sedation of Mechanically Ventilated COVID-19 Patients: Challenges and Special Considerations. Anesth Analg. 2020 Jul;131(1):e40-e41. doi: 10.1213/ANE.0000000000004887. No abstract available. PMID 32392023
- [Background] Fahy BG, Chau DF. The Technology of Processed Electroencephalogram Monitoring Devices for Assessment of Depth of Anesthesia. Anesth Analg. 2018 Jan;126(1):111-117. doi: 10.1213/ANE.0000000000002331. PMID 28786839
- [Background] Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, Chalfin DB, Masica MF, Bjerke HS, Coplin WM, Crippen DW, Fuchs BD, Kelleher RM, Marik PE, Nasraway SA Jr, Murray MJ, Peruzzi WT, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists (ASHP), American College of Chest Physicians. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002 Jan;30(1):119-41. doi: 10.1097/00003246-200201000-00020. No abstract available. PMID 11902253